CLINICAL TRIAL: NCT01633931
Title: Treatment of Adolescent Idiopathic Scoliosis Patients Using the Ellipse MAGEC System
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ellipse Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PR0038
Record Dates: First submitted 2012-07-02; First posted 2012-07-06 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect data on the use of the Ellipse MAGEC System to treat patients with adolescent idiopathic scoliosis (AIS) who have failed external brace therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Adolescent Idiopathic Scoliosis
* Failed external brace therapy defined as either (a) progression of the curve greater than 5 degrees at any time while undergoing external brace therapy, or (b) inability or unwillingness to comply with at least 16 hours per day of external bracing
* Skeletally immature (Risser Sign 0, 1, 2, or 3)
* In girls, either (a) pre-menarchal, or (b) post-menarchal by no more than 6 months
* Age between 10 and 15
* Primary Cobb angle greater than 25 degrees but not yet requiring spine fusion
* Candidate for surgical implantation of spinal instrumentation
* Patient resides locally with respect to the Investigator's clinic and is willing and able to comply with the requirements of the protocol
* Must sign informed consent to permit the use of personal health data

Exclusion Criteria:

* Patients with a pacemaker, implanted cardiac defibrillator, or any other electronic implant
* Patients who require an MRI following implantation
* Skeletally mature (Risser Sign 4 or 5; or fused tri-radiate cartilage)
* Diagnosis of other musculoskeletal or developmental illness that might be responsible for the spinal curvature
* History of previous surgical treatment for AIS

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients diagnosed with Adolescent Idiopathic Diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-03 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Change in major scoliotic curve magnitude | Change from baseline to 36 months postoperative
  Measured in degrees
Number and Types of Adverse Events | Operative through 36 months postoperative

SECONDARY OUTCOMES:
Radiographic evaluation coronal balance compared to baseline | Change from baseline to 36 months postoperative
Radiographic evaluation sagittal balance compared to baseline | Change from baseline to 36 months postoperative
Percent of patients indicated for surgical spine fusion | Change from baseline to 36 months postoperative
Quality of life assessment via SRS-30 questionnaire | Change from baseline to 36 months postoperative
Comparison of Rib Hump prominence | Change from baseline to 36 months postoperative
Expected vs. Actual Device Lengthening | All postoperative visits where lengthening is conducted

CONTACTS AND LOCATIONS:
Overall Officials: Behrooz Akbarnia, MD, Principal Investigator — San Diego Center for Spinal Disorders
Locations (1):
- University of Hong Kong, Hong Kong, Pokfulam, Hong Kong